CLINICAL TRIAL: NCT06999811
Title: Technology-Enhanced Therapy vs. Medication Monitoring for Buprenorphine Retention in Pregnant Persons
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Sara Witcraft, Research Assistant Professor-Faculty, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Pro00141060; 1K23DA062794-01 (NIH)
Record Dates: First submitted 2025-05-15; First posted 2025-05-31 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Opioid Use Disorder; Pregnancy
Keywords: Anxiety; Mental Health; Pregnancy; Psychiatry; Sleep Disorders; Substance Use; Women's Health
MeSH Terms: conditions — Opioid-Related Disorders; Anxiety Disorders; Psychological Well-Being; Sleep Wake Disorders; Substance-Related Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EMPWR (Experimental): Brief cognitive-behavioral intervention and mobile application
  Interventions: Behavioral: Empowering Pregnant Women and People Receiving medications for opioid use disorder (EMPWR)
- Control (Active Comparator): medication monitoring
  Interventions: Other: Medication monitoring (control)

INTERVENTIONS:
Behavioral: Empowering Pregnant Women and People Receiving medications for opioid use disorder (EMPWR) — EMPWR is evidence-informed, behavioral intervention to address risk factors for fear of opioid withdrawal, craving, and stress, with an adjective mobile application among pregnant women receiving opioid agonist therapies. The goal of EMPWR is to promote medication retention and adherence.
  Arms: EMPWR
Other: Medication monitoring (control) — Participants will record the dose and time buprenorphine was taken for two months via REDCap daily diaries, which will be delivered via text.
  Arms: Control

SUMMARY:
This study involves testing how useful a technology-enhanced therapy is for pregnant people prescribed buprenorphine for the treatment of opioid use disorder, compared to medication monitoring. Participants are randomized to one of the conditions. If participants are randomized to receive the therapy, participants will attend four 60-minute therapy appointments during pregnancy with an additional 30-minute therapy session towards the end of pregnancy, and 6 additional monthly postpartum (after childbirth) sessions (0-6 months postpartum). As part of the therapy program, participants will receive access to a mobile application, which will be accessible for the duration of the study. If participants are randomized to medication monitoring, participants will be asked to log each time participants take their medication for two months. All participants will also be asked to complete questionnaires at enrollment and again at 3-month postpartum and 6-months postpartum, and will be contacted randomly throughout the study to perform a medication count. The total duration of the study is between 8-12 months depending on when participants enroll (early second trimester-mid third trimester).

DETAILED DESCRIPTION:
Medication for opioid use disorder (MOUD) can effectively prevent overdose and death for pregnant and postpartum people with opioid use disorder (OUD). Yet, only half of birthing people continue to use MOUD postpartum, increasing risk for overdose two-fold. This study will evaluate feasibility of RCT methodology for a technology-enhanced behavioral intervention that aims to improve retention in and adherence to MOUD during the peripartum period compared to control (medication monitoring). The intervention contains a brief behavioral intervention targeting malleable risk factors for treatment dropout, opioid cravings, and return to illicit opioid use: anxiety sensitivity and sleep deficiency. An adjunctive mobile application will supplement therapy sessions and contains a medication adherence feature involving daily (or multiple/day) notification reminder to take medication at a scheduled time and dose consistent with the participant's prescription.

ELIGIBILITY:
Inclusion Criteria:

* currently pregnant and between 13 weeks and 0 days to 32 weeks and 6 days gestational age
* current OUD or history of OUD within past 3 years
* confirmed prescription for sublingual buprenorphine products (i.e., Suboxone, Subutex, Zubsolv) for the purpose of treating OUD
* living in the United States
* between 18-45 years of age

Exclusion Criteria:

* carrying multiples
* high-risk pregnancies including the following conditions: active hyperemesis at the time of consent or hospitalization for intractable nausea and vomiting in the current pregnancy, hypertensive disorders of pregnancy (e.g., gestational hypertension, preeclampsia), placenta previa, or vaginal bleeding in current pregnancy after the first trimester
* current psychotic symptoms and/or active suicidal intent
* experiencing cognitive or emotional impairment that precludes providing informed consent
* incarcerated/pending incarceration or institutionalized during the study period
* non-English speaking.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Pregnant people with opioid use disorder (OUD) receiving buprenorphine formulations
Enrollment: 37 (Estimated)
Dates: Start 2025-11-05 (Actual); Primary Completion 2028-10-15 (Estimated); Study Completion 2028-10-15 (Estimated)

PRIMARY OUTCOMES:
Feasibility of Recruitment | Years 3-4
  Recruitment will be assessed by the proportion of participants who agree to participate in the trial vs. total approached; success is if ≥70% of approached PPP enroll.
Retention in Active Treatment (EMPWR) | Years 3-4
  Retention will be assessed by the proportion of participants who complete 3- and 6-month postpartum follow-up assessments vs. those who prematurely terminate; success is if 70% of participants are retained for follow-up assessments.
Engagement in intervention | Years 3-4
  Overall engagement will be measured separately for the EMPWR behavioral intervention and mobile application (EMPWR condition) and daily diary completion (MM condition). To measure engagement in the EMPWR condition, we will consider it successful if 70% of participants attend all EMPWR behavioral intervention sessions, and separately, actively engage with the active components of the mobile application (i.e., 50% days logged buprenorphine, 50% assigned at-home "Practice" exercises completed). In the MM condition, we will consider completing 70% of daily diaries as successful engagement.

CONTACTS AND LOCATIONS:
Overall Officials: Sara Witcraft, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States